CLINICAL TRIAL: NCT06514157
Title: A Phase I, Open-Label, Single-dose, Single Arm Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Budesonide and Albuterol Delivered by PT027 in Healthy Chinese Participants
Brief Title: Phase I PK Study of Budesonide/Albuterol Delivered From PT027 in Healthy Chinese Participants.
Acronym: PUTUO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6935C00001
Record Dates: First submitted 2024-05-29; First posted 2024-07-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer
Keywords: Chinese healthy volunteer; Phase I
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BDA MDI (Experimental): Each randomized participant will receive a single dose of BDA MDI 160 μg/180 μg (administered as 2 actuations of 80 μg/90 μg) on Day 1 in the morning.
  Interventions: Combination Product: budesonide/albuterol sulfate metered dose inhaleor (BDA MDI)

INTERVENTIONS:
Combination Product: budesonide/albuterol sulfate metered dose inhaleor (BDA MDI) — BDA MDI 160 μg/180 μg (single dose administered as 2 actuations of 80 μg/90 μg)

SUMMARY:
A phase I study to assess the PK, safety, and tolerability of budesonide and albuterol delivered from a single dose of BDA MDI administered by inhalation in healthy Chinese participants.

DETAILED DESCRIPTION:
This is a Phase I, single centre, single arm, open-label study to gather information on the PK, safety, and tolerability of budesonide and albuterol delivered from BDA MDI after single dose administration in healthy Chinese male and female participants. Approximately 14 healthy Chinese participants, aged 18 to 55 years, will be assigned to study intervention.

The study will comprise:

A screening period of minimum 2 days and maximum 27 days Inpatient admission period during which participants will be resident from the day prior to administration of BDA MDI (Day -1) until at least 24 hours after dosing. Participants will be discharged on the morning of Day 2. The treatment will consist of a single dose of BDA MDI 160 μg/180 μg (administered as 2 actuations of 80 μg/90 μg) followed by 24 hours of plasma sampling for determination of PK parameters A Follow-up Visit within 3 to 7 days after the administration of BDA MDI.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
2. Chinese participants who are healthy
3. Body weight ≥ 45 kg for female participants and ≥ 50 kg for male participants and body BMI ≤ 26 kg/m2 at Visit 1 (screening).
4. Male and non-pregnant, non-lactating female.
5. Provision of signed and dated, written informed consent prior to any study specific procedures.
6. Resting heart rate ≥ 50 beats per minute (bpm) and ≤ 100 bpm at Visit 1 (screening) and at admission to the unit on Day -1 at Visit 2.
7. Non-smoker.
8. Must be able to demonstrate proper inhalation technique using the Vitalograph AIM device 3 repeated times as well as be able to use the BDA MDI according to instructions at Visit 1 (screening) and Day -1.

Exclusion Criteria:

1. As judged by the investigator, any evidence which in the investigator's opinion makes it undesirable for the participant to participate in the study.
2. History of any significant drug allergy or hypersensitivity to albuterol sulfate or other beta-adrenergic agonists or to budesonide or other corticosteroids.
3. Recent history of a disease or condition that would result in any residual upper respiratory airways/lung inflammatory process or residual limited lung function at the time of Day 1 at Visit 2.
4. Have any gastrointestinal, hepatic, or renal condition that might affect the absorption, distribution, biotransformation, or excretion of drugs.
5. Use of any medication within 2 weeks or within the equivalent time of 5 half-lives of taking the last dose (whichever is longer) before the study intervention, or hormonal drug products and traditional Chinese medicines within 30 days before the study intervention.
6. Participation in any other clinical investigation using an experimental drug requiring repeated blood or plasma draws within 30 days or 5 half-lives of the drugs (whichever takes longer) of Day 1 at Visit 2.
7. Have abnormal and clinically significant results on the physical examination, medical history, clinical chemistry, haematology, or urinalysis at Visit 1 (screening) or Day -1 at Visit 2.
8. Resting systolic blood pressure ≥ 140 or ≤ 90 mmHg and resting diastolic blood pressure ≥ 90 or ≤ 50 mmHg at Visit 1 (Screening) or Day -1 at Visit 2.
9. 12-lead ECG showing QTcF ≥ 450 msec for participants as indicated in the reading report assessed at Visit 1 (screening).
10. Positive test results for syphilis antibody, HBsAg, hepatitis C antibody and/or HIV I antibodies at Visit 1 (screening).
11. Have a history of alcohol or substance abuse within the previous 5 years as reported by the participant.
12. Positive results for drugs of abuse at Visit 1 (screening) or Day -1 at Visit 2.
13. Have participated in a blood/plasma donation or blood loss greater than 400 mL within 90 days, or greater than 200 mL within 30 days prior to screening (Visit 1).
14. Inability to be venipunctured or tolerate venous access as determined by the PI or designee.
15. Participants unable to give their consent, or participants of consenting age but under guardianship, or vulnerable participants.
16. In the opinion of the PI, participants who are unlikely to comply with the protocol requirements, instructions, and study-related restrictions.
17. Participants who are relatives of the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff or directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
AUClast of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration
AUCinf of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration
Cmax of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration
tmax of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration
Tlast of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration
t½λz of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration
CL/F of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration
Vz/F of budesonide and albuterol | From Day 1 pre-dose to 24 hours post dose
  To characterize the PK of budesonide and albuterol delivered from BDA MDI after single dose administration

SECONDARY OUTCOMES:
Incidence of AEs/SAEs | Screening(Day-27 to Day-2), Day-1, Day1(dosing day), Day 2, Follow-Up(Day 3 to Day7)
  To assess the safety and tolerability of budesonide and albuterol delivered from BDA MDI after single dose administration in healthy Chinese participants
Incidence of abnormal vital signs: blood pressure and pulse rate | Screening(Day-27 to Day-2), Day-1, Day1(post dose), Day 2, Follow-Up(Day 3 to Day7)
  To assess the safety and tolerability of budesonide and albuterol delivered from BDA MDI after single dose administration in healthy Chinese participants
Incidence of abnormal haematology assessments: WBC count, RBC count, Hemoglobin, Platelets and Leukocytes absolute count | Screening (Day -27 to Day -2), Day -1, Follow-up (Day 3 to Day 7)
  To assess the safety and tolerability of budesonide and albuterol delivered from BDA MDI after single dose administration in healthy Chinese participants
Incidence of abnormal 12-lead ECG parameters: heart rate, RR interval, QRS interval, PR interval, QT/QTcF interval. | Screening (Day -27 to Day -2), Day 1(post dose), Follow-up (Day 3 to Day 7)
  To assess the safety and tolerability of budesonide and albuterol delivered from BDA MDI after single dose administration in healthy Chinese participants
Incidence of abnormal clinical chemistry assessments： Sodium, potassium, calcium, urea, creatinine, ALP, ALT, AST, total bilirubin, CK albumin and fasting glucose | Screening (Day -27 to Day -2), Day -1, Follow-up (Day 3 to Day 7)
  To assess the safety and tolerability of budesonide and albuterol delivered from BDA MDI after single dose administration in healthy Chinese participants
Incidence of abnormal urinalysis： Glucose, blood, protein, microscopy(including RBC,WBC and casts) | Screening (Day -27 to Day -2), Day -1, Follow-up (Day 3 to Day 7)
  To assess the safety and tolerability of budesonide and albuterol delivered from BDA MDI after single dose administration in healthy Chinese participants

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D6935C00001_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6935C00001&attachmentIdentifier=537119f7-f115-40c7-9998-9138b52c5bcb&fileName=D6935C00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=